CLINICAL TRIAL: NCT04218604
Title: Feasibility and Efficacy of Tailoring Ablation Index to Left Atrial Wall Thickness During Atrial Fibrillation Ablation: The Ablate By-LAW Study
Brief Title: The Ablate-by-LAW Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Heart Center Leipzig - University Hospital (Other); Hospital Universitario Puerta del Mar (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Principal investigator, cardiologist, cardiac electrophysiologist, Centro Medico Teknon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ablation-by-LAW
Record Dates: First submitted 2019-12-26; First posted 2020-01-06 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter-based ablation; radiofrequency ablation; pulmonary vein isolation; left atrial wall thickness; multidetector cardiac tomography
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized AF ablation using MDCT-derived LAWT (Experimental): Pre-procedural MDCT images will be analysed in Teknon Medical Center (core-lab), using ADAS-3D™ (Galgo Medical, Barcelona, Spain) to obtain 3D atrial wall thickness maps that will be introduced into CARTO® navigation system (Biosense Webster, Diamond Bar, California, US). PVI will be performed point-by-point, aiming to complete a RF circle around the PV ostia (nephroid shape) on the 3D geometry using a ThermoCool® SmartTouch® 3.5-mm irrigated tip contact force-sensing RF ablation catheter (Biosense Webster, Inc.). AI targets will be defined by LAWT on the thickness color map, as follows: Thickness < 1 mm (red): 300; 1-2 mm (yellow): 350; 2-3 mm (green): 400; 3-4 mm (blue): 450; > 4 mm (purple): 500. The recommended power settings to reach these AI values will be, in general, 35 W for the posterior wall and 40 W for the anterior wall. Wherever local AWT is > 3 mm (green and blue colors), an increased RF power (50 W) will be permitted.
  Interventions: Procedure: Personalized atrial fibrillation ablation

INTERVENTIONS:
Procedure: Personalized atrial fibrillation ablation — Atrial fibrillation (AF) ablation adapting the ablation index (AI) target in a point-by-point manner, according the local left atrial wall thickness (LAWT), as measured by multidetector cardiac tomography (MDCT)

SUMMARY:
Of all the determinants of lesion creation during atrial fibrillation (AF) ablation, left atrial wall thickness (LAWT), as measured with multi-detector cardiac tomography (MDCT) is one key element that has been evaluated in some retrospective analyses but is not yet used per protocol to modulate the radiofrequency delivery. Adapting ablation index (AI) to LAWT would be very useful in standardising the ablation procedure with parameters fitted to every patient, enabling the development of a personalized approach that will both: i) increase efficacy by performing transmural lesions to prevent the formation of conduction gaps in the initial lesion set, and ii) increase safety by preventing excessive RF delivery on thin wall areas related to procedural complications, such as cardiac perforation or atrio-esophageal fistula. The investigators sought to evaluate the feasibility, safety, efficacy and reproducibility of guiding AF ablation procedures with the integrated MDCT-derived LAWT information.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Indication for paroxysmal atrial fibrillation ablation.
* Signed informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Previous AF ablation procedure (REDO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Arrhythmia-free survival | 1 year
  1-year atrial arrhythmia-free survival

SECONDARY OUTCOMES:
Acute procedural outcomes | 1 day
  Procedure times
Peri-procedural complications | 1 month
REDO outcomes | 2 years
  Mean LAWT at late reconnection sites

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (2):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Heart Center Leipzig University Hospital, Leipzig
- Azienda Ospedaliero-Universitaria Pisana, Pisa, Italy
- Spain (2):
  - Teknon Medical Center, Barcelona
  - Puerta del Mar University Hospital, Cadiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Alexandru Popescu B, Schotten U, Van Putte B, Vardas P. 2016 ESC Guidelines for the Management of Atrial Fibrillation Developed in Collaboration With EACTS. Rev Esp Cardiol (Engl Ed). 2017 Jan;70(1):50. doi: 10.1016/j.rec.2016.11.033. No abstract available. English, Spanish. PMID 28038729
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. J Arrhythm. 2017 Oct;33(5):369-409. doi: 10.1016/j.joa.2017.08.001. Epub 2017 Sep 15. No abstract available. PMID 29021841
- [Background] Ouyang F, Tilz R, Chun J, Schmidt B, Wissner E, Zerm T, Neven K, Kokturk B, Konstantinidou M, Metzner A, Fuernkranz A, Kuck KH. Long-term results of catheter ablation in paroxysmal atrial fibrillation: lessons from a 5-year follow-up. Circulation. 2010 Dec 7;122(23):2368-77. doi: 10.1161/CIRCULATIONAHA.110.946806. Epub 2010 Nov 22. PMID 21098450
- [Background] Cappato R, Negroni S, Pecora D, Bentivegna S, Lupo PP, Carolei A, Esposito C, Furlanello F, De Ambroggi L. Prospective assessment of late conduction recurrence across radiofrequency lesions producing electrical disconnection at the pulmonary vein ostium in patients with atrial fibrillation. Circulation. 2003 Sep 30;108(13):1599-604. doi: 10.1161/01.CIR.0000091081.19465.F1. Epub 2003 Sep 8. PMID 12963643
- [Background] Kuck KH, Hoffmann BA, Ernst S, Wegscheider K, Treszl A, Metzner A, Eckardt L, Lewalter T, Breithardt G, Willems S; Gap-AF-AFNET 1 Investigators*. Impact of Complete Versus Incomplete Circumferential Lines Around the Pulmonary Veins During Catheter Ablation of Paroxysmal Atrial Fibrillation: Results From the Gap-Atrial Fibrillation-German Atrial Fibrillation Competence Network 1 Trial. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003337. doi: 10.1161/CIRCEP.115.003337. PMID 26763226
- [Background] Ikeda A, Nakagawa H, Lambert H, Shah DC, Fonck E, Yulzari A, Sharma T, Pitha JV, Lazzara R, Jackman WM. Relationship between catheter contact force and radiofrequency lesion size and incidence of steam pop in the beating canine heart: electrogram amplitude, impedance, and electrode temperature are poor predictors of electrode-tissue contact force and lesion size. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1174-80. doi: 10.1161/CIRCEP.113.001094. Epub 2014 Nov 7. PMID 25381331
- [Background] Thiagalingam A, D'Avila A, Foley L, Guerrero JL, Lambert H, Leo G, Ruskin JN, Reddy VY. Importance of catheter contact force during irrigated radiofrequency ablation: evaluation in a porcine ex vivo model using a force-sensing catheter. J Cardiovasc Electrophysiol. 2010 Jul;21(7):806-11. doi: 10.1111/j.1540-8167.2009.01693.x. Epub 2010 Feb 1. PMID 20132400
- [Background] Barkagan M, Rottmann M, Leshem E, Shen C, Buxton AE, Anter E. Effect of Baseline Impedance on Ablation Lesion Dimensions: A Multimodality Concept Validation From Physics to Clinical Experience. Circ Arrhythm Electrophysiol. 2018 Oct;11(10):e006690. doi: 10.1161/CIRCEP.118.006690. PMID 30354405
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Natale A, Albenque JP, Kautzner J, Shah D, Michaud G, Wharton M, Harari D, Mahapatra S, Lambert H, Mansour M. Randomized, Controlled Trial of the Safety and Effectiveness of a Contact Force-Sensing Irrigated Catheter for Ablation of Paroxysmal Atrial Fibrillation: Results of the TactiCath Contact Force Ablation Catheter Study for Atrial Fibrillation (TOCCASTAR) Study. Circulation. 2015 Sep 8;132(10):907-15. doi: 10.1161/CIRCULATIONAHA.114.014092. Epub 2015 Aug 10. PMID 26260733
- [Background] Shah DC, Lambert H, Nakagawa H, Langenkamp A, Aeby N, Leo G. Area under the real-time contact force curve (force-time integral) predicts radiofrequency lesion size in an in vitro contractile model. J Cardiovasc Electrophysiol. 2010 Sep;21(9):1038-43. doi: 10.1111/j.1540-8167.2010.01750.x. PMID 20367658
- [Background] De Potter T, Van Herendael H, Balasubramaniam R, Wright M, Agarwal SC, Sanders P, Khaykin Y, Latcu DG, Maury P, Pani A, Hayes J, Kalman J, Nery P, Duncan E. Safety and long-term effectiveness of paroxysmal atrial fibrillation ablation with a contact force-sensing catheter: real-world experience from a prospective, multicentre observational cohort registry. Europace. 2018 Nov 1;20(FI_3):f410-f418. doi: 10.1093/europace/eux290. PMID 29315382
- [Background] Ho SY, Cabrera JA, Tran VH, Farre J, Anderson RH, Sanchez-Quintana D. Architecture of the pulmonary veins: relevance to radiofrequency ablation. Heart. 2001 Sep;86(3):265-70. doi: 10.1136/heart.86.3.265. PMID 11514476
- [Background] Ho SY, Sanchez-Quintana D. The importance of atrial structure and fibers. Clin Anat. 2009 Jan;22(1):52-63. doi: 10.1002/ca.20634. PMID 18470938
- [Background] Kistler PM, Ho SY, Rajappan K, Morper M, Harris S, Abrams D, Sporton SC, Schilling RJ. Electrophysiologic and anatomic characterization of sites resistant to electrical isolation during circumferential pulmonary vein ablation for atrial fibrillation: a prospective study. J Cardiovasc Electrophysiol. 2007 Dec;18(12):1282-8. doi: 10.1111/j.1540-8167.2007.00981.x. Epub 2007 Oct 3. PMID 17916142
- [Background] Takahashi K, Okumura Y, Watanabe I, Nagashima K, Sonoda K, Sasaki N, Kogawa R, Iso K, Ohkubo K, Nakai T, Hirayama A. Relation Between Left Atrial Wall Thickness in Patients with Atrial Fibrillation and Intracardiac Electrogram Characteristics and ATP-Provoked Dormant Pulmonary Vein Conduction. J Cardiovasc Electrophysiol. 2015 Jun;26(6):597-605. doi: 10.1111/jce.12660. Epub 2015 May 1. PMID 25777254
- [Background] Suenari K, Nakano Y, Hirai Y, Ogi H, Oda N, Makita Y, Ueda S, Kajihara K, Tokuyama T, Motoda C, Fujiwara M, Chayama K, Kihara Y. Left atrial thickness under the catheter ablation lines in patients with paroxysmal atrial fibrillation: insights from 64-slice multidetector computed tomography. Heart Vessels. 2013 May;28(3):360-8. doi: 10.1007/s00380-012-0253-6. Epub 2012 Apr 22. PMID 22526381
- [Background] Nakamura K, Funabashi N, Uehara M, Ueda M, Murayama T, Takaoka H, Komuro I. Left atrial wall thickness in paroxysmal atrial fibrillation by multislice-CT is initial marker of structural remodeling and predictor of transition from paroxysmal to chronic form. Int J Cardiol. 2011 Apr 14;148(2):139-47. doi: 10.1016/j.ijcard.2009.10.032. Epub 2009 Nov 10. PMID 19906452
- [Background] Chikata A, Kato T, Sakagami S, Kato C, Saeki T, Kawai K, Takashima S, Murai H, Usui S, Furusho H, Kaneko S, Takamura M. Optimal Force-Time Integral for Pulmonary Vein Isolation According to Anatomical Wall Thickness Under the Ablation Line. J Am Heart Assoc. 2016 Mar 15;5(3):e003155. doi: 10.1161/JAHA.115.003155. PMID 27068636
- [Background] Sun JY, Yun CH, Mok GSP, Liu YH, Hung CL, Wu TH, Alaiti MA, Eck BL, Fares A, Bezerra HG. Left Atrium Wall-mapping Application for Wall Thickness Visualisation. Sci Rep. 2018 Mar 8;8(1):4169. doi: 10.1038/s41598-018-22089-z. PMID 29520005
- [Background] Bishop M, Rajani R, Plank G, Gaddum N, Carr-White G, Wright M, O'Neill M, Niederer S. Three-dimensional atrial wall thickness maps to inform catheter ablation procedures for atrial fibrillation. Europace. 2016 Mar;18(3):376-83. doi: 10.1093/europace/euv073. Epub 2015 Apr 4. PMID 25842272
- [Background] Schaeffer B, Willems S, Sultan A, Hoffmann BA, Luker J, Schreiber D, Akbulak R, Moser J, Kuklik P, Steven D. Loss of Pace Capture on the Ablation Line During Pulmonary Vein Isolation versus "Dormant Conduction": Is Adenosine Expendable? J Cardiovasc Electrophysiol. 2015 Oct;26(10):1075-80. doi: 10.1111/jce.12759. Epub 2015 Aug 29. PMID 26183341
- [Result] Das M, Loveday JJ, Wynn GJ, Gomes S, Saeed Y, Bonnett LJ, Waktare JEP, Todd DM, Hall MCS, Snowdon RL, Modi S, Gupta D. Ablation index, a novel marker of ablation lesion quality: prediction of pulmonary vein reconnection at repeat electrophysiology study and regional differences in target values. Europace. 2017 May 1;19(5):775-783. doi: 10.1093/europace/euw105. PMID 27247002
- [Result] Hussein A, Das M, Chaturvedi V, Asfour IK, Daryanani N, Morgan M, Ronayne C, Shaw M, Snowdon R, Gupta D. Prospective use of Ablation Index targets improves clinical outcomes following ablation for atrial fibrillation. J Cardiovasc Electrophysiol. 2017 Sep;28(9):1037-1047. doi: 10.1111/jce.13281. Epub 2017 Jul 26. PMID 28639728
- [Result] Taghji P, El Haddad M, Phlips T, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Evaluation of a Strategy Aiming to Enclose the Pulmonary Veins With Contiguous and Optimized Radiofrequency Lesions in Paroxysmal Atrial Fibrillation: A Pilot Study. JACC Clin Electrophysiol. 2018 Jan;4(1):99-108. doi: 10.1016/j.jacep.2017.06.023. Epub 2017 Sep 27. PMID 29600792
- [Result] Inoue J, Skanes AC, Gula LJ, Drangova M. Effect of Left Atrial Wall Thickness on Radiofrequency Ablation Success. J Cardiovasc Electrophysiol. 2016 Nov;27(11):1298-1303. doi: 10.1111/jce.13065. Epub 2016 Sep 16. PMID 27510229
- [Result] Pambrun T, Combes S, Sousa P, Bloa ML, El Bouazzaoui R, Grand-Larrieu D, Thompson N, Martin R, Combes N, Boveda S, Haissaguerre M, Albenque JP. Contact-force guided single-catheter approach for pulmonary vein isolation: Feasibility, outcomes, and cost-effectiveness. Heart Rhythm. 2017 Mar;14(3):331-338. doi: 10.1016/j.hrthm.2016.12.008. Epub 2016 Dec 7. PMID 27940124
- [Result] Steven D, Reddy VY, Inada K, Roberts-Thomson KC, Seiler J, Stevenson WG, Michaud GF. Loss of pace capture on the ablation line: a new marker for complete radiofrequency lesions to achieve pulmonary vein isolation. Heart Rhythm. 2010 Mar;7(3):323-30. doi: 10.1016/j.hrthm.2009.11.011. Epub 2009 Nov 12. PMID 20185104
- [Result] Eitel C, Hindricks G, Sommer P, Gaspar T, Kircher S, Wetzel U, Dagres N, Esato M, Bollmann A, Husser D, Hilbert S, Zaker-Shahrak R, Arya A, Piorkowski C. Circumferential pulmonary vein isolation and linear left atrial ablation as a single-catheter technique to achieve bidirectional conduction block: the pace-and-ablate approach. Heart Rhythm. 2010;7(2):157-64. doi: 10.1016/j.hrthm.2009.10.003. Epub 2009 Oct 12. PMID 20036199
- [Derived] Alderete J, Fernandez-Armenta J, Zucchelli G, Sommer P, Nazarian S, Falasconi G, Soto-Iglesias D, Silva E, Mazzocchetti L, Bergau L, Khoshknab M, Penela D, Berruezo A. The Ablate-by-LAWT multicentre prospective study: Personalized paroxysmal atrial fibrillation ablation with ablation index adapted to local left atrial wall thickness. J Interv Card Electrophysiol. 2024 Dec;67(9):2089-2099. doi: 10.1007/s10840-024-01871-2. Epub 2024 Jul 15. PMID 39009785

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT04218604/Prot_SAP_ICF_002.pdf